CLINICAL TRIAL: NCT06443099
Title: The Effect of Cold Needle and Shotblocker on Pain and Satisfaction in Intramuscular Injection Pain: A Randomized Controlled Trial
Brief Title: Needle and Shotblocker on Pain and Satisfaction in Intramuscular Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Doctor of Teaching Member, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Shotblocker
Record Dates: First submitted 2024-05-29; First posted 2024-06-05 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Intramuscular Injection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- shotblocker group (Experimental): It is a C-shaped plastic tool with small blunt protrusions on one side that contact the skin. It does not have any side effects. The protruding surface of the ShotBlocker is pressed against the skin during injection and the injection is performed through the opening. It is thought to provide pain control as an application of gate control theory. In addition to the IM injection application procedure, after the skin is cleaned in the patient group, the protruding part of the ShotBlocker (Bionix, Press Firmly, USA) will be placed in contact with the skin. The ShotBlocker will be pressed firmly against the skin and the injection will be made through the central opening of the ShotBlocker. Once the injection is complete, the ShotBlocker will be removed from the skin.
  Interventions: Other: Different methods used after intramuscular injection
- Cold needle group (Experimental): In addition to the IM injection procedure, a cold needle tip will be used in the needle tip changing procedure step. For this, before the application, the 25 Gauge orange syringe tip will be placed in a cold thermos and kept at 0-2 degrees Celsius with ice batteries. The appropriate temperature range will be checked with a digital thermometer.
  Interventions: Other: Different methods used after intramuscular injection
- Control group (No Intervention): Applications will be carried out according to the IM injection application protocol. Identifying the deltoid region. Clean the area around the injection site (five cm) with 70% disposable alcohol cotton in circular motions, wait for the alcohol to dry in the area (5 seconds). Injecting the drug every 10 sec/ml. 10 seconds before withdrawing the needle. wait. Retracting the needle straight and steady at the angle at which the tissue was entered.

INTERVENTIONS:
Other: Different methods used after intramuscular injection — Different methods will be used during intramuscular injection. One of them is shotblocker. There are studies reporting that it reduces pain according to the gate control theory. The other method is cold injection. In this method, the injector tips will be cooled to 0-2 degrees and used in injection application.
  Arms: Cold needle group; shotblocker group

SUMMARY:
In this study, it is aimed to compare cold needle and shotblocker in intramuscular injection pain. This is a triple-blind randomized clinical trial. June September 2024, the universe of the research will be composed of patients who applied to the emergency department of Necmettin Erbakan University Faculty of Medicine Hospital for cyanocobalamin injection. Considering that losses may occur during the data collection process, the study will be completed with a total of 120 patients. Intramuscular injection of the deltoid November will be applied to the intervention-1 group with a cold needle, intervention-2 group with a shotblocker, and the control group with the standard method. People will be determined by block randomization. After each application, the pain and satisfaction due to the injection will be evaluated. The data will be compared between the groups.

DETAILED DESCRIPTION:
This study aims to compare cold injection and ShotBlocker in intramuscular injection pain. This is a triple-blind randomized clinical trial. The population of the research will consist of patients who applied to the emergency department of Necmettin Erbakan University Faculty of Medicine Hospital to receive cyanocobalamin injection between June and September 2024. Considering that losses may occur during the data collection process, the study will be completed with a total of 120 patients. The data of the study will be collected with the "Patient Diagnosis Form", "Visual Analog Scale (VAS)" and "Injection Satisfaction Scale". Block randomization method will be used to assign participants to groups. All injections will be performed by a single nurse working in the injection unit in accordance with the research procedure. Once the injection procedure is completed, participants will be asked to rate injection pain and satisfaction. Pain assessment will be performed by another emergency nurse who is independent from the study and contributes to the study. Researchers will participate in this process as observers. The people who will perform the application and evaluate the pain and satisfaction will be different. In this way, the person evaluating the pain will not know which application was performed on the participant, and blinding will be ensured. Additionally, the data of the study will be coded as A, B and C and entered into SPSS, thus ensuring statistical blinding. Thus, it is planned to conduct the research with triple blinding. All injections will be made using cyanocobalamin injection (1 ml), 5 cc syringe, 25 Gauge orange syringe tip. Before the injection, it will be checked whether the pain score is "0" with VAS. The participant will be given a Fowler position, the deltoid area will be checked on the arm to be treated, the arm will be flexed and brought closer to the body, and the position will be given. Injections will be given to each group according to the IM injection application protocol. Intramuscular injection will be applied to the deltoid muscle in the intervention-1 group, with a cold needle, in the intervention-2 group, with a shot blocker, and in the control group, with the standard method. Subjects will be determined by block randomization. All participants will be allowed to rest for two minutes after each injection. After two minutes, they will be asked to mark the level of pain caused by the procedure on the VAS. Similarly, they will be asked to mark their satisfaction with the procedure on the injection satisfaction scale. Then, the line marked by the person will be measured with a 10 cm ruler and the numerical equivalent of pain and satisfaction will be determined. Data will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* No problems with speaking and understanding Turkish,
* Body mass index (BMI) between 18.5 and 30,
* Just starting the first dose of cyanocobalamin treatment,
* No history of allergy to the drug,
* No vision, hearing or perception problems,
* Having orientation to place and time,
* No sensorimotor deficit,
* No history of diabetes,
* Not taking oral or parenteral analgesic treatment before the application,
* VAS score before injection is "0",
* No deficiency in limbs,
* No pregnancy,
* Female individuals who are not in their menstrual cycle,
* Volunteering to participate in the research.

Exclusion Criteria:

* Another injection into the deltoid area,
* Development of drug-related allergy or other complications,
* Scar, incision, infection, sensitivity, burn, cut, etc. in the injection area. to be found,
* Wants to leave the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
injection pain | up to 2 months
  Visual Pain Scale (Visual Analog Scale-VAS) is a reliable measurement tool developed to measure individuals' pain levels. The scale is simple, interesting, quick to fill out, and easy to score. There are subjective descriptive expressions at both ends of a 10-cm ruler (0: lowest pain level and 10: highest pain level). The patient will be asked to mark the place on the line that expresses his/her pain.

SECONDARY OUTCOMES:
injection satisfaction | up to 2 months
  The injection satisfaction scale is a 0-10 cm ruler that will be used to evaluate patients' satisfaction with the injection application. Patients will mark their satisfaction with the injection application on the ruler.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)